CLINICAL TRIAL: NCT02605694
Title: A Phase 2, Randomized Study of Duvelisib Administered in Combination With Rituximab vs R-CHOP in Subjects With Relapsed/Refractory Follicular Lymphoma (FRESCO)
Brief Title: Duvelisib With Rituximab vs R-CHOP in Subjects With Relapsed/Refractory Follicular Lymphoma (FRESCO)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is focusing on studies which can enable registration of duvelisib
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-21; 2015-004729-15 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-16 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — duvelisib; Rituximab; R-CHOP protocol; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Duvelisib 25 mg will be administered orally twice daily (BID) during 21-day cycles (Cycles 1-6) followed by 28-day cycles (Cycle 7 and beyond) until disease progression or unacceptable toxicity; and Rituximab (375 mg/m2) will be administered as an intravenous (IV) infusion on Day 1 of Cycles 1-6 (21-day cycles).
  Interventions: Drug: Duvelisib; Drug: Rituximab
- Arm 2 (Active Comparator): R-CHOP will be administered as follows:
  IV infusion on Day 1 of Cycles 1-6 (21-day cycles)
  * Cyclophosphamide (750 mg/m2)
  * Doxorubicin hydrochloride (50 mg/m2)
  * Vincristine sulfate (1.4 mg/m2) (2 mg maximum)
  * Rituximab (375 mg/m2) Orally on Days 1-5 of Cycles 1-6 (21-day cycles)
  * Prednisone (100 mg) will be administered.
  Interventions: Drug: Rituximab; Drug: R-CHOP; Drug: Prednisone

INTERVENTIONS:
Drug: Duvelisib — 25 mg will be administered orally twice daily (BID) during 21-day cycles (Cycles 1-6) followed by 28-day cycles (Cycle 7 and beyond) until disease progression or unacceptable toxicity
  Other Names: IPI-145
  Arms: Arm 1
Drug: Rituximab — 375 mg/m2 will be administered as an intravenous (IV) infusion on Day 1 of Cycles 1-6 (21-day cycles).
  Other Names: MabThera; Rituxan
Drug: R-CHOP — IV infusion on Day 1 of Cycles 1-6 (21-day cycles)
  * Cyclophosphamide (750 mg/m2)
  * Doxorubicin hydrochloride (50 mg/m2)
  * Vincristine sulfate (1.4 mg/m2) (2 mg maximum)
  * Rituximab (375 mg/m2)
  Other Names: Rituximab; CHOP
  Arms: Arm 2
Drug: Prednisone — 100 mg orally on Days 1-5 of Cycles 1-6 (21-day cycles)
  Other Names: Deltasone
  Arms: Arm 2

SUMMARY:
Phase II study to evaluate the efficacy and safety of DR vs R-CHOP in subjects with relapsed/refractory FL

DETAILED DESCRIPTION:
This is a phase 2, randomized, two-arm, open-label study designed to evaluate the efficacy and safety of Duvelisib Administered in Combination with Rituximab vs R-CHOP in Subjects with Relapsed/Refractory Follicular Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of FL: Grade 1, 2, or 3a
2. Progressed within 24 months of initiating an alkylator-based chemotherapy regimen given as either first- or second-line therapy; single-agent chlorambucil therapy does not fulfill this requirement Note: subjects must have received at least 2 cycles of alkylator-based chemotherapy to be eligible
3. Previously received rituximab, either as single agent or as part of any combination regimen, and also meet one of the following requirements:

   1. Progressed within 24 months of initiating alkylator-based chemotherapy in the first line and received no additional anticancer therapy
   2. Progressed within 24 months of initiating alkylator-based chemotherapy in the first line and subsequently progressed within 24 months of receiving any second-line treatment and received no additional anticancer therapy
   3. Progressed within 24 months of initiating alkylator-based chemotherapy in the second line and received no additional anticancer therapy
4. Appropriate to receive R-CHOP
5. At least 1 measurable disease lesion > 1.5 cm in at least one dimension by computed tomography (CT), CT-PET, or magnetic resonance imaging (MRI)
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (corresponds to Karnofsky Performance Status [(KPS) ≥60%])
7. For women of childbearing potential (WCBP): negative serum β human chorionic gonadotropin (βhCG) pregnancy test within 1 week before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 12 consecutive months for women >55 years of age)

Exclusion Criteria:

1. Clinical evidence of transformation to a more aggressive subtype of lymphoma or grade 3B FL
2. Received ≥ 3 previous anticancer regimens prior to enrollment
3. Received prior R-CHOP therapy
4. Previous receipt of any anthracycline
5. Contraindication to any of the individual components of CHOP (cyclophosphamide, vincristine, doxorubicin and prednisone) Severe allergic or anaphylactic reaction to any monoclonal antibody therapy, murine protein, or known hypersensitivity to any of the study drugs
6. Received prior allogeneic transplant
7. Received prior treatment with a phosphoinositide-3-kinase (PI3K) inhibitor
8. History of tuberculosis treatment within the two years prior to randomization
9. History of chronic liver disease, veno-occlusive disease, alcohol abuse
10. Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids >20 mg of prednisone (or equivalent) QD
11. Ongoing treatment for systemic bacterial, fungal, or viral infection at screening
12. Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A (CYP3A)
13. Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
14. Concurrent active malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix
15. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or a pacemaker within the last 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Time from randomization to documented disease progression, or death due to any cause, whatever comes first, assessed up to approximately 44 months.
  Progression Free Survival (PFS), defined according to the revised International Working Group (IWG) criteria as assessed by the Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Every 3-6 Cycles (Cycles 1-6 are 21-days; after Cycle 7 are 28-days) from randomization until first documented progression. Subjects will be evaluated for progression or the primary analysis of PFS, whichever occurs first.
  Complete Response Rate (CRR) with complete response defined according to the revised IWG criteria as assessed by the IRC
Overall Response Rate (ORR) | Every 3-6 Cycles (Cycles 1-6 are 21-days; after Cycle 7 are 28-days) from randomization until first documented progression or the primary analysis of PFS, whichever occurs first.
  ORR defined as best response of complete response (CR) or partial response/remission (PR), according to the revised IWG criteria as assessed by the IRC
Overall Survival | Every 6 months until the primary analysis for PFS or 3 years from randomization, whichever occurs later.
Safety (Treatment Emergent Adverse Events (TEAEs) and changes in safety laboratory values as assessed by NCI-CTCAE, version 4.03) | Continuous from informed consent until 30 days from last dose
  Adverse events (AEs) and abnormal laboratory values
Pharmacokinetics: Evaluate the Duvelisib concentration in plasma sample | Cycle 1 Day 15, Cycle 2 Day 1 and 15 (Cycles 1-6 are 21-day cycles)
  Evaluate the Duvelisib concentration in plasma sample
Duration of Response | Every 3-6 Cycles (Cycles 1-6 are 21-days; after Cycle 7 are 28-days) from the first documented response to first documented progression or death, whichever occurs first.
  DOR defined as the time from the first documented response to the first documentation of progressive disease (PD) according to the revised IWG criteria or death due to any cause (for subjects with CR or PR only)
Pharmacokinetics: Evaluate IPI-656 (metabolite) concentration in plasma sample | Cycle 1 Day 15, Cycle 2 Day 1 and 15 (Cycles 1-6 are 21-day cycles)
  Evaluate IPI-656 (metabolite) concentration in plasma sample

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- Miami, Florida, United States